CLINICAL TRIAL: NCT03964363
Title: Pre-operative Physical Training for Elderly Patients with Frailty
Brief Title: Home-based Prehabilitation for Elderly Patients
Acronym: TRAilty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: PV5951
Record Dates: First submitted 2019-04-28; First posted 2019-05-28 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Frail Elderly Syndrome
Keywords: Frailty; preoperative period; surgery; breathing exercise; postoperative complications; resistance training; endurance training; anaesthesia; activities of daily living; patient reported outcome; prehabilitation; perioperative care; elderly; prevention
MeSH Terms: conditions — Frailty; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: This trail is designed as a prospective, multicentre, randomized controlled study with two parallel groups with a total of four arms. Patients with a scheduled elective surgery will be randomly assigned into treatment and control group after having been screened for frailty. A subgroup will be formed by patients who will receive a transcatheter aortic valve implantation (TAVI). The preventative effect of a behaviour modification will subsequently be compared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Prehabilitation (Experimental): Participants are scheduled for elective surgery and follow the home-based prehabilitation for 11-17 days
  Interventions: Behavioral: Unsupervised home-based physical prehabilitation
- Prehabilitation + TAVI (Experimental): Study participants who will undergo a TAVI form a subgroup with a modified enrolment procedure and longer duration of the intervention. The prehabilitation period is extended to 30 days.
  Interventions: Behavioral: Unsupervised home-based physical prehabilitation
- Control (No Intervention): Participants are initially evaluated for frailty prior to scheduled surgery but subsequently receive regular care without a prehabilitation program. All pre- and postsurgical evaluations will be identical to the prehabilitation group.
- Control+TAVI (No Intervention): The subgroup of participants who undergo a TAVI will be compared to a group of patients who will have had the same procedure. Hence the control group will also receive a screening via phone but then receive regular care. Follow-up after surgery will be identical in all groups.

INTERVENTIONS:
Behavioral: Unsupervised home-based physical prehabilitation — Subsequent to screening and initial testing for frailty syndrome, participants receive an information booklet containing a selection of exercises, which allows independent prehabilitation at home.
  Arms: Prehabilitation; Prehabilitation + TAVI

SUMMARY:
As a consequence of the increasing life expectancy hospitals are seeing a growing number of elderly patients undergoing elective surgery. These patients are likely to suffer from one or more chronic illnesses, malnutrition, reduced physical strength and mobility and sensory impairment. Age related loss of resilience in combination with these conditions often results in frailty. Frailty syndrome describes a reduction in weight, mobility and strength, as well as declining cognitive capacities and reduced performance in daily life activities. This decline in constitution is accompanied by an increased risk of complications and mortality in the period after surgery. Frail patients are generally admitted to hospital for a longer period and are readmitted more often.

A multitude of studies has demonstrated that these risks can be significantly reduced by offering frail patients a prevention program prior to their surgery. These prevention programs are often referred to as prehabilitation and combine strength and cardiovascular training with breathing exercises. Despite the obvious benefits, prehabilitation programs are not yet commonly applied outside of research settings as they carry considerable costs and required additional skilled personnel.

In response to the unmet need for a widely applicable, cost and personnel efficient prehabilitation program a home-based prehabilitation program has been designed. This prehabilitation allows patients to safely perform an individualised set of exercises without relying on a personal trainer or a training group. Efficiency and feasibility will be evaluated in this study.

DETAILED DESCRIPTION:
The average age of hospital patients has steadily increased with the demographic change of Germany's ageing population. In 2014, more than 27 million people living in Germany were older than 60 years and more than one third of this group had to undergo surgery within that year.

A relevant proportion of this patient group has to be considered frail or pre-frail. Over a lifetime every individual experiences a physiological reduction of functional capacity across all organ systems resulting in frailty. Consequently, physical and psychological stress, such as a hospital stay and surgery cannot be readily compensated. Therefore, frailty is a highly predictive pre-operative risk factor for increased post-operative morbidly and mortality, prolonged hospital stay and loss of independence. Multiple studies have demonstrated post-operative outcome of frail patients can be drastically improved if these patients are identified prior to elective surgery and enrolled in a multimodal prehabilitation program. The core of prehabilitation is physical exercise next to nutritional and psychological support. The improvement of cardiovascular condition, ventilator capacity and muscle strength gained during prehabilitation resulted in a reduced incidence of complications including pneumonia, shorter hospital stays and improved quality of life. Yet despite these benefits prehabilitation is not yet widely available outside of clinical studies as they carry considerable costs and demand additional skilled personnel.

In order to provide prehabilitation to a larger group of patients, a pre-operative exercise program was developed, that can safely be followed by pre-frail and frail patients at home without the need of continuous instruction and supervision by a trainer or physiotherapist. Efficacy and feasibility will be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

* pre-frail or frail according to (Longitudinal Urban Cohort Ageing Study) LUCAS-functional index
* scheduled for elective surgery
* planned ward admission for at least 24h after surgery

Exclusion Criteria:

* Refusal of participation
* Presentation less than 2 weeks prior to scheduled procedure
* Pre-existing pronounced immobility (wheelchair bound, paresis of both arms or both legs)
* Minor surgical interventions such as small excisions of superficial tissues, small interventions for haemorrhoids, curettage, gastroscopy

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 512 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-10-12 (Actual)

PRIMARY OUTCOMES:
Quality of recovery: QoR-15 | 7 days postoperative
  The quality of recovery after surgery and anaesthesia is measured using the QoR-15 questionnaire. The resulting score indicates self-reported patent well-being and perceived support with higher scores (0-100) indicating a better quality of recovery. (8)

SECONDARY OUTCOMES:
Quality of recovery: QoR-15 | 3 months postoperative
  The quality of recovery after surgery and anaesthesia is measured using the QoR-15 questionnaire. The resulting score indicates self-reported patent well-being and perceived support with higher scores (0-100) indicating a better quality of recovery. (8)
Health related quality of life: Questionnaire Short Form-12 (SF-12) | preoperative, 3 months postoperative
  The World Health Organisation Disability Assessment Schedule (WHODAS) assesses six domains of functioning relating to the quality of life. Quality of life is measured using the Questionnaire Short Form-12 (SF-12), which indicates physical and psychological wellbeing. Higher scores indicate a better health related quality of life.
Activities of daily living | preoperative, 7 days and 3 months postoperative
  The Lawton-Brody Instrumental Activities of Daily Living is used to assess the ability to perform activities that are central to living independently. A lower score indicates better functioning. The score ranges between 8 - 31
Cognitive performance | preoperative, 7 days and 3 months postoperative
  Cognitive functioning will be tested with the Montreal Cognitive assessment (MOCA), a standardised test that includes memory recall, verbal fluency and visuospatial abilities. A total score between 0 and 30 is calculated with a higher score indicating better cognitive functioning.
Mobility | preoperative, 3 months postoperative
  The time up&go-test, in which the subject starts from a sitting position, walks a defined distance of 3 m and returns to a sitting position on a chair is indicative of fall risk and mobility. The chosen cut-off in this study is 10 seconds.
Muscle strength | preoperative, 7 days postoperative
  Grip strength is widely used in the diagnosis of frailty and sarcopenia. It will be measured with a hand held dynamometer in kg, using the dominant hand if possible.
Incidence of postoperative complications | preoperative, 7 days and 3 months postoperative
  Complications reported in hospital files or patient interview
Duration of hospital admission | 3 months postoperative
  Day of admission to day of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Olotu, MD, Principal Investigator — Department of Anaesthesiology, University Medical Center Eppendorf
Locations (3):
- Germany (3):
  - Rotkreuzklinikium München, München, Bavaria
  - University Medical Center Eppendorf, Hamburg, Hamburg
  - Agaplesion Diakonieklinikum Hamburg, Hamburg, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim SW, Han HS, Jung HW, Kim KI, Hwang DW, Kang SB, Kim CH. Multidimensional frailty score for the prediction of postoperative mortality risk. JAMA Surg. 2014 Jul;149(7):633-40. doi: 10.1001/jamasurg.2014.241. PMID 24804971
- [Background] Makary MA, Segev DL, Pronovost PJ, Syin D, Bandeen-Roche K, Patel P, Takenaga R, Devgan L, Holzmueller CG, Tian J, Fried LP. Frailty as a predictor of surgical outcomes in older patients. J Am Coll Surg. 2010 Jun;210(6):901-8. doi: 10.1016/j.jamcollsurg.2010.01.028. Epub 2010 Apr 28. PMID 20510798
- [Background] Jadczak AD, Makwana N, Luscombe-Marsh N, Visvanathan R, Schultz TJ. Effectiveness of exercise interventions on physical function in community-dwelling frail older people: an umbrella review of systematic reviews. JBI Database System Rev Implement Rep. 2018 Mar;16(3):752-775. doi: 10.11124/JBISRIR-2017-003551. PMID 29521871
- [Background] Boden I, Skinner EH, Browning L, Reeve J, Anderson L, Hill C, Robertson IK, Story D, Denehy L. Preoperative physiotherapy for the prevention of respiratory complications after upper abdominal surgery: pragmatic, double blinded, multicentre randomised controlled trial. BMJ. 2018 Jan 24;360:j5916. doi: 10.1136/bmj.j5916. PMID 29367198
- [Background] Beggs T, Sepehri A, Szwajcer A, Tangri N, Arora RC. Frailty and perioperative outcomes: a narrative review. Can J Anaesth. 2015 Feb;62(2):143-57. doi: 10.1007/s12630-014-0273-z. Epub 2014 Nov 25. PMID 25420470
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725
- [Background] Jammer I, Wickboldt N, Sander M, Smith A, Schultz MJ, Pelosi P, Leva B, Rhodes A, Hoeft A, Walder B, Chew MS, Pearse RM; European Society of Anaesthesiology (ESA) and the European Society of Intensive Care Medicine (ESICM); European Society of Anaesthesiology; European Society of Intensive Care Medicine. Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine: European Perioperative Clinical Outcome (EPCO) definitions: a statement from the ESA-ESICM joint taskforce on perioperative outcome measures. Eur J Anaesthesiol. 2015 Feb;32(2):88-105. doi: 10.1097/EJA.0000000000000118. PMID 25058504